CLINICAL TRIAL: NCT00343941
Title: A Phase II Multicentre, Randomized, Double Blind, Parallel Group, Placebo Controlled Pilot Study of Tucaresol at Two Dosing Levels (25,50 mg) in HIV-1 Infected Adult Subjects With Plasma HIV-1 RNA < 50 Copies/ml on Stable Highly Active Antiretroviral Therapy Regimen for at Least 3 Months
Brief Title: Tucaresol As Add-On To HAART (Highly Active Antiretroviral Therapy) In Chronic HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100438
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infection
Keywords: HIV-1 infection; Tucaresol; Viral suppression
MeSH Terms: conditions — HIV Infections | interventions — tucaresol

INTERVENTIONS:
Drug: Tucaresol tablets 25 mg

SUMMARY:
This is a pilot study designed to determine a dose and schedule of Tucaresol that can be administered to HIV-1 infected subjects on HAART (highly active antiretroviral therapy) with viral suppression without occurrence of significant adverse events and that results in significant changes in cell mediated immunity.

ELIGIBILITY:
Inclusion Criteria:

* Currently on licensed triple combination therapy, which is defined as two nucleoside analogues (2 NRTI) (excluding Abacavir) and a protease inhibitor (PI) (including boosted PI regimens) or non nucleoside reverse transcriptase inhibitor (NNRTI).
* Must be on the same treatment for at least 3 months prior to study without plans to alter therapy for the next 3 months.

Plasma HIV-1 RNA (ribonucleic acid)< 50 copies/mL at screening with a documented history of continuous suppression defined as: the last two readings < 50 copies/mL for a period of at least 3 months prior to screening.

* Documented CD4+ lymphocyte cell count =350 cells/ml at screening with at least one reading =350 cells/mL in the preceding 3 months and CD4 nadir >200 cells/ml.

HBsAg (human hepatitis B Virus surface antigen) and HCV-Ab (human hepatitis C Virus antibody) negative.

Exclusion Criteria:

* History of hyperimmune or allergic reactions to drug treatment within 3 months prior to study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45
Dates: Start 2004-11

PRIMARY OUTCOMES:
Significant increase from baseline in IFN-g (Interferon gamma) EliSpot cellular responses at day 70 following peptide stimulation of PBMC (peripheral blood monocytic cells) of subjects after the second dosing cycle of study drug (days 56 to 62).

SECONDARY OUTCOMES:
Proportion of subjects developing drug related and treatment-limiting Adverse Events leading to discontinuation of study drug during the period of study and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (6):
- Italy (6):
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto